CLINICAL TRIAL: NCT04327635
Title: Safety Evaluation of Intracoronary Infusion of Extracellular Vesicles in Patients Following Coronary Stent Implantation (EV-CSI)
Brief Title: Safety Evaluation of Intracoronary Infusion of Extracellular Vesicles in Patients Following Coronary Stent Implantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Christopher J. McLeod (Other)
Collaborators: Rion LLC (Unknown)
Responsible Party: Sponsor-Investigator, Christopher J. McLeod, Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 18-011636
Record Dates: First submitted 2020-03-25; First posted 2020-03-31 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Percutaneous Coronary Intervention
Keywords: Coronary Stent Placement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PEP in Coronary Stent Implantation (Experimental): Patients undergoing a percutaneous coronary intervention (PCI) and possible stent placement procedure will receive a one-time intracoronary infusion of PEP within 20 minutes after stent placement or post-dilation (whichever comes last).
  Interventions: Drug: PEP

INTERVENTIONS:
Drug: PEP — A biological drug made of certain parts of blood from living blood donors obtained from a certified blood bank. At the time of cardiac catheterization patients will undergo one-time intracoronary infusion of 10 milliliters of PEP dosage consisting of approximately 5%, 10%, or 20% PEP. PEP dose will be infused immediately distal to the newly placed stent over approximately 5 minutes.

SUMMARY:
The purpose of this study is to determine the safety of using a biological drug called PEP in people who have had a coronary stent placed. A biological drug is a substance that is made from a living organism or its products (parts). In this case, PEP is made of certain parts of blood from living blood donors obtained from a certified blood bank. PEP comes in a powder form and is mixed with heparinized saline (a solution used to prevent clots in catheters) to create a solution that can be injected. The investigators want to see if PEP can be used to stop or slow heart damage.

DETAILED DESCRIPTION:
Patients who undergo Percutaneous Coronary Intervention (PCI) will be treated with a single dose of PEP within 20 minutes after stent placement or post-dilation (whichever is last). Subjects will be screened at the time of emergency room presentation. Subjects will be treated in the cardiac catheterization laboratory where the PCI will be completed and PEP will be administered. Subjects will be followed for one year after PEP administration through clinic visits.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing ≥1 elective, urgent, or emergent coronary stent implantation
* Angiographic evidence of TIMI 3 flow through the stented vessel after stent placement
* Angiographic evidence of residual stenosis visually <30% after stent placement
* Willing and able to provide signed informed consent
* Lives within 90 mile radius of study site
* Willing and able to return to study site for all follow-up visits

Exclusion Criteria:

* Prior solid organ transplantation at any time
* Pregnant or lactating at screening
* Known presence of chronic systemic inflammatory disorder that requires ongoing therapy with immunosuppressive agents
* Known immune system compromise including but not limited to human immunodeficiency virus (HIV), hepatitis A, hepatitis B (HBV) or hepatitis C (HCV) infection
* Known history of malignancy of any type except non-melanoma skin cancer
* Known serum creatinine >2 mg/dL or GFR ≤30 mL/min within the last twelve months
* Known AST, ALT, and/or bilirubin (total) elevated twice the upper limit of normal for age & gender within the last twelve months
* Known Hemoglobin lower than 8.0 g/dL within the last twelve months
* Known current illicit drug use at screening
* Other major surgical procedure or major trauma within the previous 14 days prior to enrollment
* Female of child bearing potential who is unwilling to agree to use acceptable contraception methods for 3 months after receiving the investigational drug
* Pacemaker/ICD implant in place
* Adult lacking decision-making capacity
* Prisoner
* Non-English speaking
* English-speaking but illiterate
* Legally blind
* Known allergy to heparin or heparin-induced thrombocytopenia
* Known history of positive SARS-CoV2 testing within the last 30 days
* DNR/DNI status prior to PCI procedure or planned DNR/DNI status after PCI procedure
* Homeless or no permanent address at the time of enrollment

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2025-10-22 (Actual); Study Completion 2025-10-22 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLTs) and maximum tolerated dose (MTD) of a single dose (10 mL) of PEP at escalating concentrations of extracellular vesicles delivered at a single time point (after PCI). | Days 1-14 of the study period for each study participant.
  DLTs are defined as: signs of infection present in the judgement of a reviewing MD, CTCAE Grade 2 or higher bronchial stricture (rhonchi/wheezing), or CTCAE Grade 3 or higher defined as new or reoccurring angina or anginal equivalent after infusion with PEP; elevated ALT, AST, total or direct bilirubin, unless due to procedural complications or complications of ischemic cardiomyopathy (ICM); decreased hemoglobin or platelet level, unless due to procedural complications or complications of ICM; sustained ventricular arrhythmia during PEP infusion; hypersensitivity or anaphylaxis during PEP infusion; any other grade 3 or higher adverse event.

SECONDARY OUTCOMES:
Infarction scar size | Day 7 and Day 40 of the study period for each study participant.
  Cardiac MRI will be used to assess myocardial infarction scar size.
Ejection fraction | Day 7 and Day 40 of the study period for each study participant.
  Cardiac MRI will be used to assess ejection fraction.
Alloimmune Response | Day 1 (Baseline/Screening) visit, Day 40 and Day 365
  Class I & II Antibody Single Antigen Bead testing will be completed. Changes will be documented and evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Guy S Reeder, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD, related data dictionaries, and all IPD that underlie results in a publication available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Prior to study initiation, the study protocol and informed consent form will be provided to Rion, LLC. During the study, all safety reports (as they happen or quarterly), and all SAEs as they happen will be reported to Rion, LLC. At the end of the study after database is locked, a formal clinical study report will be provided to Rion, LLC.
Access Criteria: IPD will only be shared with the collaborator, Rion, LLC.

REFERENCES:
- [Derived] Kisby CK, Shadrin IY, Peng LT, Stalboerger PG, Trabuco EC, Behfar A, Occhino JA. Impact of Repeat Dosing and Mesh Exposure Chronicity on Exosome-Induced Vaginal Tissue Regeneration in a Porcine Mesh Exposure Model. Female Pelvic Med Reconstr Surg. 2021 Mar 1;27(3):195-201. doi: 10.1097/SPV.0000000000001017. PMID 33620904